CLINICAL TRIAL: NCT05836675
Title: Effects of an Intradialytic Exercise Program on Quality of Life, Sexual Function, and Sexual Satisfaction of Patients Undergoing Hemodialysis
Brief Title: Quality of Life and Sexual Life in Hemodialysis Patients: Effects of an Intradialytic Exercise Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autónoma de Yucatán (Other)
Responsible Party: Principal Investigator, Adriana Cruz-Bañares, PhD Student, Universidad Autónoma de Yucatán
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Fmed-05-23
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Chronic Kidney Diseases; Sexual Dysfunction
Keywords: Intradialytic exercise; Hemodialysis; Sexual Dysfunctions; Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Sexual Dysfunction, Physiological; Kidney Diseases | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: There will be one single group that will act as their own control throughout the intervention
Masking Description: Since it is an exercise intervention, the participants cannot be masked. When the analysis and interpretation of the data is preformed, the investigator will not know the participants identification data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental Intradialytic exercise (Experimental): Aerobic, resistance and Kegel exercises
  Interventions: Other: Intradialytic exercise

INTERVENTIONS:
Other: Intradialytic exercise — The exercise program will be carried out during dialysis time. Participants will be asked to carry out cycling for 15-20 minutes, resistance exercises, and Kegel exercises during the first 2 hours of their regular routine hemodialysis session. Exercise can be done with rest periods as necessary.
  Other Names: Exercise

SUMMARY:
The aim of the study is to investigate whether an intradialytic exercise program can improve the quality of life, sexual function, and sexual satisfaction in patients undergoing hemodialysis.

DETAILED DESCRIPTION:
When diagnosed with Chronic Kidney Disease phase 5, patients are dialyzed to remove waste products and toxins from the blood that kidneys can´t longer filter. Although hemodialysis removes most of the toxins and allows health improvement, patients continue reporting a low quality of life and limitations in their functional independence.

Within the context of quality of life, sexuality is an important factor; a high incidence of sexual dysfunctions has been reported among hemodialysis patients. Although poorly addressed, it impacts family and couple relationships, emotions, and mental health.

Exercise interventions improve physical function and quality of life, and since some of the mechanisms involved in exercise are also involved in sexual activity, an exercise intervention could be an effective approach to sexual dysfunctions without the risk and stigma of sexual or drug therapy.

Therefore the study aims to implement an intradialytic exercise program involving aerobic, resistance, and Kegel exercises (specific to the pelvic floor) and determine its effects on quality of life, sexual function, and sexual satisfaction in patients undergoing hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Participants with stage 5 of Chronic Kidney Disease
* Participants that are undergoing hemodialysis for at least 3 months
* Participants between 18 and 70 years old
* Their participation is voluntary and they have signed the informed consent form
* Participants that have medical approval from their nephrologist

Exclusion Criteria:

* Participants with severe cardiovascular damage (NYHA >3)
* Participants with a high probability of receiving a transplant within 6 months
* Participants with psychiatric or psychological disorders such as severe depression (Beck Index) that can affect their ability to consent or participate in the study
* Participants that perform physical exercise at least 2 times a week for the last 3 months or more
* Participants with bilateral lower limb amputation
* Participants with vascular access located in lower limbs
* Pregnant participants

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2023-08-08 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2025-06-19 (Actual)

PRIMARY OUTCOMES:
Kidney Disease and Quality of life | 6 months
  This outcome will be measured by means of the Kidney Disease and Quality of life Questionnaire (KDQOL-SF36) which is a specific questionnaire designed for patients with kidney disease on dialysis; it was developed by the Kidney Disease Quality of life Working Group as a self-report measure of health-related quality of life perceived by patients with this condition. It is a self-reported questionnaire that includes generic items for chronic conditions (SF-36) and disease-specific items. The minimum score is 0 and the maximum score is 100; a higher score means a better quality of life.
Sexual Function | 6 months
  For men, the outcome will be measured by means of the International Index of Erectile Function (IIEF) which is a questionnaire designed to evaluate erectile dysfunction. It was developed with the aim of assessing the effects of the Sildenafil clinical trial and is now the gold standard measure for erectile dysfunction. It is a self-reported questionnaire that includes 15 questions regarding erectile function, orgasm function, sexual arousal and satisfaction. The minimum score is 5 and the maximum score is 75; a higher score means less dysfunction while a lower one means a more severe dysfunction.
  For women, the outcome will be measured by means of the Female Sexual Function Index (FSFI) which is a questionnaire designed to assess female sexual function. It is a self-reported inventory with 19 questions addressing desire, arousal, lubrication, orgasm, satisfaction and pain. An score under 26 expresses the presence of a dysfunction.
Sexual Satisfaction | 6 months
  This outcome will be measured by means of the New Sexual Satisfaction Scale (NSSS) which is a questionnaire designed to measure global sexual satisfaction regardless gender, sexual orientation or relationship status. It is a self-reported questionnaire that includes 20 questions regarding sexual sensations, sexual awareness, sexual exchange, emotional connection and sexual activity. The maximum score is 100; a higher score means a better perception of their sexual satisfaction.

SECONDARY OUTCOMES:
Depression and anxiety | 6 months
  This will be measured by means of the Beck Depression and Anxiety Scale. It is a sef-reported questionnaire that assesses the clinical symptoms present in depression, it is commonly used to assess the severity of the disease. It consists in 21 questions that ask about how the individual has felt in the past 2 weeks. The minimum score is 0 and the maximum one is 63; a highest score means a more severe depression.
Body Image Perception | 6 months
  This outcome will be measured by means of a Body Image Perception Questionnaire designed to assess the level of body image disturbance in patients undergoing dialysis or with kidney transplant. It is a self-reported questionnaire with 20 questions with a minimum of 0 points and a maximum of 80; a higher score means a more severe body image disturbance.
Functional Capacity-6mwt | 6 months
  The functional capacity will be measured by means of the 6-minute-walk-test (6mwt) which is defined as a constant load stress test that measures the distance the participant can walk in a period of 6 minutes, at a fast pace and with possible resting breaks. The test is widely used in chronic kidney disease patients and reflects the functional ability to perform daily activities.
Functional Capacity-STS30 | 6 months
  The functional capacity will also be measured by means of the sit-to-stand test (STS30) which assesses the lower limb function by asking the participant to sit and stand as fast as possible as many times in 30 seconds.
Functional Capacity-HandgripTest | 6 months
  The functional capacity will also be measured by means of the Handgrip Test which assesses the upper limb muscle strength by performing a dynamometry. The participant will squizz the grip until they reach their maximum strength for 2 seconds, the test will be performed twice.

CONTACTS AND LOCATIONS:
Overall Officials: Héctor A Rubio-Zapata, Dr, Study Director — Universidad Autónoma de Yucatán; Adriana Cruz-Bañares, Principal Investigator — Universidad Autónoma de Yucatán
Locations (2):
- Mexico (2):
  - Hospital Regional de Alta Especialidad de la Península de Yucatán, Mérida, Yucatán
  - Unidad Médica de Atención Ambulatoria del Instituto Mexicano del Seguro Social, Mérida, Yucatán

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salehi F, Mangolian Shahrbabaki P, Dehghan M, Amirihosseini M. Can passive pedaling improve sexual function in patients under hemodialysis? A randomized clinical trial. Ther Apher Dial. 2022 Feb;26(1):130-139. doi: 10.1111/1744-9987.13691. Epub 2021 Jun 11. PMID 34032376